CLINICAL TRIAL: NCT04176029
Title: Point of Care Lung Ultrasound to Differentiate Causes of Respiratory Distress in Children With Severe Malaria
Brief Title: Lung Ultrasound in Children With Severe Malaria
Acronym: LUSiSM
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); University of Kinshasa (Other)
Responsible Party: Sponsor
Other Study IDs: MAL19008
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-01

CONDITIONS: Severe Malaria
Keywords: severe malaria; lung ultrasound; prevalence of pulmonary diagnoses
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children admitted with confirmed severe malaria
  Interventions: Device: lung ultrasound

INTERVENTIONS:
Device: lung ultrasound — Lung ultrasound is performed using an 12-regions technique i.e. six areas on each side of the chest, two ventral, two lateral and two posterior. The lung ultrasound examination is estimated to take around 10 minutes of time.

SUMMARY:
A prospective cohort study, with 171 children admitted for severe malaria that will be included in the cohort. The study will take place in Kinshasa, Democratic Republic of Congo.

The primary objective is to evaluate the prevalence of five pre-specified pulmonary diagnoses that can be facilitated by the use of LUS (normal lung or acidotic breathing, ARDS, concomitant pneumonia, hydrostatic pulmonary oedema, pleural effusion).

DETAILED DESCRIPTION:
A prospective cohort study, with 171 children (between 1 - 14 years) admitted for severe malaria that will be included in the cohort. The study will take place at the Maluku District Hospital, located in Kinshasa, Democratic Republic of Congo.

Lung ultrasound will be performed on admission, h24, and unscheduled timepoints (in case of respiratory deterioration during hospital stay). Lung auscultation and peripheral capillary oxygen saturation (SpO2) will be assessed at each time points. All children will be observed from admission to hospital discharge. At 30 days a phone call will be made by the study staff to follow up clinical conditions of the child.

The total duration for each subject's participation in the study is approximately 1 month. The study period is approximately 12 months

Funder: The Wellcome Trust (ITPA grant) WT-iTP-2019/005

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 and 14 years;
* Admitted for confirmed severe malaria (i.e. positive peripheral blood slide for malaria parasite and/or positive rapid diagnostic test for malaria in combination with one or more clinical or laboratory severity criteria detailed below).
* Informed consent signed

Clinical features of severe malaria

* Cerebral malaria; A Glasgow Coma Scale of less than 11 or a Blantyre coma scale less than 3 in preverbal children
* Respiratory distress (costal indrawing, use of accessory muscles, nasal flaring, deep breathing or severe tachypnea (respiratory rate > upper normal limit for age)
* Jaundice (visible jaundice)
* Circulatory collapse or shock: age <12 systolic blood pressure < 70mm Hg; age > 12 systolic blood pressure <80mm Hg with cool extremities or capillary refill time >3 seconds
* Spontaneous bleeding
* Multiple generalized convulsions: more than two episodes within 24h
* Prostration, i.e. generalized weakness so that the patient is unable to sit, stand or walk without assistance

Laboratory features and other findings

* Metabolic acidosis (venous plasma bicarbonate < 15mmol/l or base excess < -2.2mEq/L)
* Severe anaemia (age <12: hematocrit < 15% or haemoglobin < 5g/dl; age>12: hematocrit < 20% or hemoglobin < 7 g /dl)
* Hypoglycaemia (< 2.2mmol/l or < 40mg/dl)
* Hyperparasitaemia defined as > 10%
* Hyperlactataemia (venous lactate < 5 mmol/L)
* Kidney dysfunction (blood urea >20mmol/L)

Exclusion Criteria:

* Co-morbidity which, in the judgement of the investigator or treating physician, would place the subject at undue risk or interfere with the patient's treatment or results of the study. E.g. immediate transfer needed.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children admitted for severe malaria
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion of children diagnoses | On the day of hospital admission
  Proportion of children diagnosed with (1) respiratory distress with normal lungs (acidosis) in the first 6 hours after hospital admission, (2) concomitant pneumonia, (3) hydrostatic pulmonary oedema, (4) pleural effusion and (5) acute respiratory distress syndrome (ARDS).

SECONDARY OUTCOMES:
Proportion of children that fulfill the criteria for a new pulmonary diagnosis >6 hours from admission. | From admission to discharge, aproximately 1 week
  Proportion of children without respiratory symptoms and a normal lung on lung ultrasound on admission that fulfil the criteria for a new pulmonary diagnosis >6h from admission.
Median lung ultrasound score | On the day of hospital admission
  Median lung ultrasound score (range 0 to 36) on the first lung ultrasound performed after admission.
Percentage agreement between a positive lung auscultation (bilateral crepitations) and a lung ultrasound consistent with pulmonary oedema. | From hospital admission to discharge, aproximately 1 week
  Percentage agreement between a positive lung auscultation (bilateral crepitations) and a lung ultrasound consistent with pulmonary oedema.
Hospital mortality and 30 days mortality | On hospital discharge, maximum 30 days after admission to hospital
  Mortality rate in children with severe malaria suffering from a pulmonary complication at admission or during hospitalization and 30 day follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- The Maluku District Hospital, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of MORU. With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy. (http://www.tropmedres.ac/data-sharing-policy)